CLINICAL TRIAL: NCT02092922
Title: A Phase 2 Trial of Filanesib in Relapsed/Refractory Multiple Myeloma (AfFIRM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-520-215; 2014-001051-23 (EudraCT Number); C4371002 (Other: Pfizer)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Advanced Multiple Myeloma
MeSH Terms: interventions — filanesib; KIF11 protein, human; Filgrastim; Granulocyte Colony-Stimulating Factor; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filanesib (Experimental)
  Interventions: Drug: Filanesib, KSP (Eg5) inhibitor; intravenous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous

INTERVENTIONS:
Drug: Filanesib, KSP (Eg5) inhibitor; intravenous — multiple dose, single schedule
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — standard of care

SUMMARY:
The AfFIRM Study is a Phase 2 study during which patients with advanced multiple myeloma will receive single-agent investigational study drug filanesib (ARRY-520). Patients will be followed to determine the effectiveness of filanesib in treating myeloma. Approximately 160 patients from North America and Europe will be enrolled in this study.

Eligible patients will have received at least two prior lines of therapy; have received prior bortezomib and lenalidomide; and have disease refractory to carfilzomib and/or pomalidomide.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with confirmed multiple myeloma whose treatment history must include all of the following:

  1. Received at least 2 prior lines of therapy (induction therapy and stem cell transplant ± maintenance are to be considered a single line of therapy).
  2. Received at least 2 cycles of a bortezomib-containing regimen and 2 cycles of a lenalidomide-containing regimen, unless intolerant to these agents (defined as requiring discontinuation due to toxicity).
  3. Disease refractory to a carfilzomib-containing regimen and/or a pomalidomide containing regimen. Refractory is defined as either failure to achieve a minimal response (MR) or better while on therapy, or development of progressive disease (PD) while on therapy or within 60 days from last dose of therapy.
* Measurable multiple myeloma disease, defined as meeting at least one of the following criteria within 14 days prior to first dose of study drug:

  1. A monoclonal Ig (M-protein) concentration on serum protein electrophoresis (SPEP) of ≥ 1.0 g/dL.
  2. Measurable urinary light chain secretion by quantitative analysis using urine protein electrophoresis (UPEP) of ≥ 200 mg/24 hours.
  3. Involved serum free light chain (FLC) level ≥ 10 mg/dL, provided the serum FLC ratio is abnormal.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 within 14 days prior to first dose of study drug.
* Adequate hematology, hepatic and renal function laboratory values within 14 days prior to first dose of study drug.
* Additional criteria exist.

Key Exclusion Criteria:

* Prior treatment with filanesib (ARRY-520) or any other KSP inhibitor.
* Past or current plasma cell leukemia.
* Primary amyloidosis (amyloidosis associated with multiple myeloma is allowed).
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes).
* Autologous or allogeneic stem cell or bone marrow transplant within 3 months prior to first dose of study drug.
* Concomitant malignancies or previous malignancies (other than multiple myeloma) with less than a 2-year disease-free interval at the time of first dose of study drug. Patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or Stage 1 prostate cancer are eligible irrespective of the time of diagnosis.
* Use of an investigational agent that is not expected to be cleared by the time of first dose of study drug or that has been demonstrated to have prolonged side effects. Patients must have recovered from all side effects to a Grade 0 or 1 (except alopecia and neuropathy).
* Any severe concurrent disease or condition (including severe graft-versus-host disease, requirement for dialysis, symptomatic congestive heart failure [New York Heart Association Class III or IV], unstable angina pectoris, cardiac arrhythmia) which, in the judgment of the Investigator, would make the patient inappropriate for study participation.
* Known positive serology for the human immunodeficiency virus (HIV), active hepatitis B and/or hepatitis C.
* Acute active infection requiring treatment.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
In patients with low Baseline alpha 1-acid glycoprotein (AAG), assess the efficacy of the study drug in terms of objective response rate. | up to 2 years

SECONDARY OUTCOMES:
In patients with high Baseline AAG, assess the efficacy of the study drug in terms of objective response rate. | up to 2 years
In all patients, assess the efficacy of the study drug in terms of duration of response. | up to 2 years
In all patients, assess the efficacy of the study drug in terms of progression-free survival. | up to 2 years
In all patients, assess the efficacy of study drug in terms of overall survival. | up to 2 years
In all patients, assess the safety of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | up to 2 years
In a subset of all patients, characterize the pharmacokinetics (PK) of the study drug in terms of plasma concentration-time profiles. | 6 months
In a subset of all patients, assess the correlation between study drug exposure and changes in corrected QT interval (QTc) in terms of changes in QTc versus time-matched study drug plasma concentrations. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (29):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Hematology Oncology, P.C., Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Mount Sinai Medical Center, New York, New York
  - NY Presbyterian - Weill Cornell Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Cancer Care Northwest, Spokane Valley, Washington
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Jewish General Hospital, Montreal, Quebec
- France (8):
  - Centre Hospitalier Lyon-Sud, Bierre-Benite Cedex
  - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU Hotel Dieu, Nantes
  - G.H.U Caremeau, Nîmes
  - Institut Universitaire de Cancer, Toulouse
  - CHU tours-Hopital Bretonneau, Tours
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - TU Dresden Medizinische Fakultat, Medizinische Klinik und Poliklinik I, Dresden
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - University of Tubingen, Tübingen
  - Julius Maximilians Universitat Wurzburg, Würzburg
- Greece (2):
  - General Hospital of Athens "Evangelismos", Athens
  - University of Athens School of Medicine, Athens
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Quiron de Zaragoza, Zaragoza
- United Kingdom (5):
  - Barts Health NHS Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - Southhampton General Hospital, Southhampton
  - The Royal Marsden NHS Foundation Trust, Surrey
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests